CLINICAL TRIAL: NCT01751360
Title: SYR-472 Open-label Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: SYR-472/OCT-002; U1111-1137-2768 (Registry Identifier: UTN (WHO)); JapicCTI-122024 (Registry Identifier: JapicCTI (Japan))
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — trelagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SYR-472 100mg (Experimental): SYR-472 100mg
  Interventions: Drug: SYR-472

INTERVENTIONS:
Drug: SYR-472

SUMMARY:
To evaluate the efficacy and safety of treatment with SYR-472 in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

-1. The participant is judged to be capable of understanding and complying with protocol requirements by the investigator or subinvestigator.

2. The participant can sign and date a written, informed consent form prior to the initiation of any study procedures.

Exclusion Criteria:

-1. The participant has concurrent serious cardiac disease, serious cerebrovascular disorder, or serious pancreatic or hematological disease

. 2. The participant is assessed to be ineligible for the study by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2013-08-01 (Actual); Study Completion 2013-08-01 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 7 days
  Blood Glucose

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda (Note: This product was divested to Teijin Pharma Limited in 2023)
Locations (1):
- Suita-shi, Osaka, Japan